CLINICAL TRIAL: NCT06554951
Title: Study of Extracellular Vesicles (EV) in Patients Undergoing CAR-T Cell Therapy
Brief Title: Study of Extracellular Vesicles (EV) in Patients Undergoing CAR-T Cell Therapies
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Francesca Bonifazi, MD, Head of Program of Advanced Cellular Therapies, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: CARE_24
Record Dates: First submitted 2024-08-09; First posted 2024-08-15 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: CAR-T Cell Therapy; Extracellular Vesicles
MeSH Terms: interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Patients who are candidates for CAR-T cell therapy for hematologic malignancy — This study will include patients who undergo CAR-T cell infusion at participating centers during the 18-month duration of the enrollment period. A total of 100 patients are expected to be enrolled, including 80 patients for the prospective part and 20 for the retrospective part.

SUMMARY:
Patients with refractory/relapse hematologic oncology disease may benefit from innovative therapy such as Car-T cells. Factors strongly predictive of outcome and response are unknown. Extracellular vesicles are recognized as a mode of intercellular communication and are reminiscent of the cell of origin. They are currently candidates to be biomarkers for this biomarker of phenomena occurring in tissues. The working hypothesis is that they may be predictive of outcome and toxicity, as some preliminary data have suggested.

Therefore, the aim of the study concerns I dentification of potential CAR-EV biomarkers associated with neurological toxicity after infusion of CAR-T cells.

ELIGIBILITY:
Inclusion Criteria:

* patients affeccted by any hematological malignancies (r/r B cell lymphoma, B cell acute leukemia and multiple myeloma) undergoing (or whit indication to) CAR-T cell infusion with a CAR-T cell product;
* age: 18 years or greater;
* obtained written consent to the study participation.

Exclusion Criteria:

* none

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include all patients who will undergo to CAR-T cell infusion per any hematological malignancies with AIFA approved CAR-T cell product.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-31 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Response rate to treatment with CAR-T cells | 18 months
  For lymphoma: complete remission is defined by the absence of signs, symptoms, and PET/CT of the disease as described by Mac Manus MP et al. Cancer Imaging. 2007;7:10-8 For multiple myeloma: complete remission is defined as absence of M protein signs using standard tests, disappearance of any soft tissue plasmacytomas, and less than 5% plasma cells in bone marrow aspirates (Fernandez de Larrea C et al. Biol Blood Marrow Transplant. 2011 Jul;17:1084-7).
  For acute leukemia: complete remission is defined with less than 5% blasts in os-seo marrow and all other blood cell counts have returned to normal levels.Dohner H et al Blood. 2022;140:1345-1377.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes